CLINICAL TRIAL: NCT00571025
Title: Genetic Risk Assessment and Counseling for Alzheimer's Disease
Brief Title: Risk Evaluation and Education for Alzheimer's Disease
Acronym: REVEAL I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Robert C. Green, MD, MPH, Boston University School of Medicine
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IA0126; 5R01HG002213 (NIH)
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer's Disease
Keywords: Mild Cognitive Impairment; disease/disorder proneness/risk; family genetics; genetic counseling; genetic marker; genetic polymorphism; genetic susceptibility
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Disease Susceptibility; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): AD risk assessment based on family history and APOE genotype
  Interventions: Behavioral: APOE Disclosure
- 2 (Active Comparator): AD risk assessment based on family history alone
  Interventions: Behavioral: APOE Disclosure

INTERVENTIONS:
Behavioral: APOE Disclosure — Individuals are provided with a lifetime percentage risk of developing Alzheimer's disease and told their own APOE genotype.

SUMMARY:
The purpose of this study is to determine the characteristics of those who obtain genetic susceptibility testing for Alzheimer's disease with APOE disclosure and to study the psychological and behavioral consequences of providing this information.

DETAILED DESCRIPTION:
Advances in genetic research have led to an increased number of testing procedures to determine future risk of disease among at-risk individuals. An increasing number of genes are being identified that confer susceptibility for a given disease rather than inevitably causing it. Given that such genes may provide risk information for common diseases (e.g., stroke, depression), there is a growing need to understand how at-risk populations might respond to the option of genetic susceptibility testing. A prominent case in point is Alzheimer's disease (AD).

Participation in this study requires an initial phone call which will elicit some medical and family history information about the participant. A first in-person visit to the clinic will consist of an education session and the administration of some tests to assess memory and thinking skills. This visit will take approximately 2-3 hours. Approximately 2 weeks later, participants will return to have their blood drawn for genetic testing. Participants will then be randomized to one of two groups. Those in the experimental arm will receive information on their risk based on their family history and APOE genotype, while those in the active comparator arm will receive information on their risk for developing Alzheimer's disease based on their family history alone. Participants will be followed for 1 year following disclosure of results with 2 additional clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult children of a person with clinically diagnosed and/or autopsy-confirmed Alzheimer's disease
* 18 years or older

Exclusion Criteria:

* Current dementia
* Current untreated depression

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2000-08; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiological Studies-Depression Scale (CES-D) | baseline, 6 weeks, 6 months, 12 months post-disclosure
Beck Anxiety Inventory (BAI) | baseline, 6 weeks, 6 months, 12 months post-disclosure

SECONDARY OUTCOMES:
Impact of Events Scale (IES) | 6 weeks, 6 months, 12 months post-disclosure
Future Attitudes Scale (FAS) | baseline, 6 weeks, 6 months, 12 months post-disclosure
Positive and Negative Affect Schedule (PANAS) | baseline, 6 weeks, 6 months, 12 months post-disclosure

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Green, MD, MPH, Principal Investigator — Boston University
Locations (3):
- United States (3):
  - Boston University School of Medicine, Boston, Massachusetts
  - Weill Medical College of Cornell University, New York, New York
  - Case Western Reserve University, Cleveland, Ohio

REFERENCES:
- [Background] Farrer LA, Cupples LA, Haines JL, Hyman B, Kukull WA, Mayeux R, Myers RH, Pericak-Vance MA, Risch N, van Duijn CM. Effects of age, sex, and ethnicity on the association between apolipoprotein E genotype and Alzheimer disease. A meta-analysis. APOE and Alzheimer Disease Meta Analysis Consortium. JAMA. 1997 Oct 22-29;278(16):1349-56. PMID 9343467
- [Background] Green RC, Clarke VC, Thompson NJ, Woodard JL, Letz R. Early detection of Alzheimer disease: methods, markers, and misgivings. Alzheimer Dis Assoc Disord. 1997;11 Suppl 5:S1-5; discussion S37-9. doi: 10.1016/s0197-4580(96)80334-4. PMID 9348421
- [Background] Green RC, Cupples LA, Go R, Benke KS, Edeki T, Griffith PA, Williams M, Hipps Y, Graff-Radford N, Bachman D, Farrer LA; MIRAGE Study Group. Risk of dementia among white and African American relatives of patients with Alzheimer disease. JAMA. 2002 Jan 16;287(3):329-36. doi: 10.1001/jama.287.3.329. PMID 11790212
- [Derived] Green RC, Roberts JS, Cupples LA, Relkin NR, Whitehouse PJ, Brown T, Eckert SL, Butson M, Sadovnick AD, Quaid KA, Chen C, Cook-Deegan R, Farrer LA; REVEAL Study Group. Disclosure of APOE genotype for risk of Alzheimer's disease. N Engl J Med. 2009 Jul 16;361(3):245-54. doi: 10.1056/NEJMoa0809578. PMID 19605829